CLINICAL TRIAL: NCT02182076
Title: Safety and Pharmacokinetics/Bioavailability of a Single Dose of 150 mg BIBF 1120 Administered as Soft Gelatine Capsules With and Without Food to Healthy Male Volunteers in an Open, Randomised, Intra-individual Crossover Comparison Design
Brief Title: Pharmacokinetics/Bioavailability of BIBF 1120 Administered to Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1199.17
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — nintedanib

ARMS (2):
- fasted administration of BIBF 1120 (Active Comparator): 150 mg of BIBF 1120 ES soft gelatine capsules in fasting state
  Interventions: Drug: BIBF 1120
- fed administration of BIBF 1120 (Experimental): three 50 mg BIBF 1120 soft gelatine capsule immediately after a high fat, high caloric meal
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — 150 mg of BIBF 1120 ES soft gelatine capsules

SUMMARY:
Study to assess pharmacokinetics and the extend of absorption of a single dose of BIBF 1120 soft gelatine capsule with food effect (BA) in healthy subjects respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with GCP (Good Clinical Practice) and local legislation
* Age ≥21 and ≤55 years
* Body Mass Index ≥18.5 kg/m2 and ≤29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders
* History of orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* History of any bleeding disorder including prolonged or habitual bleeding, other hematologic disease or cerebral bleeding (e.g. after a car accident)or commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* Female gender
* Male subjects must agree to minimize the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or a medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intra-uterine device, tubal ligation, hormonal contraceptive since at least two months and diaphragm with spermicide

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-10; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve in plasma over time from zero time extrapolated to infinity) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
Cmax (maximum observed concentration in plasma) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug

SECONDARY OUTCOMES:
tmax (time from dosing to reach Cmax) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
t1/2 (terminal half-life in plasma) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
MRTpo (mean residence time in the body) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
CL/F (apparent clearance in plasma following extravascular administration) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
Vz/F (apparent volume of distribution during the terminal phase following extravascular administration) | Pre-dose and 15, 30, 45 min, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 33, 48 hours after each administration of study drug
Incidence and intensity of adverse events | up to 14 days
Changes from baseline in vital signs (systolic and diastolic blood pressure, Pulse rate) | up to 14 days
Changes from baseline in laboratory tests | up to 14 days
Assessment of global tolerability on a 4-point scale | Day 3 of each treatment period
Changes from baseline in 12-lead electrocardiogram | up to 14 days